CLINICAL TRIAL: NCT00785239
Title: CryoSpray Ablation(tm)Thoracic Patient Registry
Status: Withdrawn | Type: Observational
Why Stopped: Business Reasons
Sponsor: CSA Medical, Inc. (Industry)
Collaborators: Reset Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-00031
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Lung Cancer; Emphysema; Chronic Bronchitis; COPD; Asthma; Sarcoidosis; Mesothelioma
Keywords: Malignant Airway Disease; Benign Airway Disease; Lung Cancer; Emphysema; Chronic Bronchitis; COPD; Asthma; Sarcoidosis; Mesothelioma; CryoSpray Ablation; Cryotherapy; Cryospray; Cryo
MeSH Terms: conditions — Lung Neoplasms; Emphysema; Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive; Asthma; Sarcoidosis; Mesothelioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to create a patient registry to collect and analyze information on subjects treated with the CryoSpray Ablation™ System post-510K approval.

DETAILED DESCRIPTION:
The proposed registry is a prospective, multi-center study of patients that are currently undergoing CryoSpray Ablation™. A maximum of 50 investigational sites will participate in this study.

The study population consists of patients who are being treated with the CryoSpray Ablation™ System for thoracic diseases. Enrolled subjects must have a signed consent form for data collection.

ELIGIBILITY:
Inclusion Criteria:

Patients who are being treated with the CryoSpray Ablation™ System for lung and for thoracic diseases.

Exclusion Criteria:

* Subjects with thoracic or airway obstructions and diseases who were not treated with the CryoSpray Ablation™ System.
* Subjects under the age of 18 years.
* Subjects unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of subjects treated with the CryoSpray Ablation™ System in the airway or for thoracic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Primary objectives of the study are to enable analysis of patient outcomes 2 years following final treatment and estimate the effectiveness of the device in eradicating, decreasing and downgrading of the diseases. | 2 years post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: William Krimsky, M.D., Principal Investigator — Franklin Square Hospital Center

REFERENCES:
- [Background] Johnston MH, Eastone JA, Horwhat JD, Cartledge J, Mathews JS, Foggy JR. Cryoablation of Barrett's esophagus: a pilot study. Gastrointest Endosc. 2005 Dec;62(6):842-8. doi: 10.1016/j.gie.2005.05.008. PMID 16301023
- [Background] Johnston CM, Schoenfeld LP, Mysore JV, Dubois A. Endoscopic spray cryotherapy: a new technique for mucosal ablation in the esophagus. Gastrointest Endosc. 1999 Jul;50(1):86-92. doi: 10.1016/s0016-5107(99)70352-4. PMID 10385730
- [Background] Ell C, May A, Gossner L, Pech O, Gunter E, Mayer G, Henrich R, Vieth M, Muller H, Seitz G, Stolte M. Endoscopic mucosal resection of early cancer and high-grade dysplasia in Barrett's esophagus. Gastroenterology. 2000 Apr;118(4):670-7. doi: 10.1016/s0016-5085(00)70136-3. PMID 10734018
- [Background] Champion G, Richter JE, Vaezi MF, Singh S, Alexander R. Duodenogastroesophageal reflux: relationship to pH and importance in Barrett's esophagus. Gastroenterology. 1994 Sep;107(3):747-54. doi: 10.1016/0016-5085(94)90123-6. PMID 8076761
- [Background] Eisen GM, Sandler RS, Murray S, Gottfried M. The relationship between gastroesophageal reflux disease and its complications with Barrett's esophagus. Am J Gastroenterol. 1997 Jan;92(1):27-31. PMID 8995932
- [Background] Johnston MH. Cryotherapy and other newer techniques. Gastrointest Endosc Clin N Am. 2003 Jul;13(3):491-504. doi: 10.1016/s1052-5157(03)00044-8. PMID 14629105
- [Background] Cash BD, Johnston LR, Johnston MH. Cryospray ablation (CSA) in the palliative treatment of squamous cell carcinoma of the esophagus. World J Surg Oncol. 2007 Mar 16;5:34. doi: 10.1186/1477-7819-5-34. PMID 17367523
- [Background] Pinsonneault C, Fortier J, Donati F. Tracheal resection and reconstruction. Can J Anaesth. 1999 May;46(5 Pt 1):439-55. doi: 10.1007/BF03012943. PMID 10349923
- [Background] Field JK, Youngson JH. The Liverpool Lung Project: a molecular epidemiological study of early lung cancer detection. Eur Respir J. 2002 Aug;20(2):464-79. doi: 10.1183/09031936.02.00290202. PMID 12212983